CLINICAL TRIAL: NCT06736509
Title: An Open-Label Study to Assess the Long-term Safety of AXS-05 in Subjects With Dementia of the Alzheimer's Type, ADVANCE-2 and ACCORD-2 Extension Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study AXS-05-AD-305 was terminated due to completion of overall program objectives.
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXS-05-AD-305
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type; Alzheimer Disease; Agitation, Psychomotor
Keywords: AD Agitation; AXS-05; NMDA receptor antagonist; dextromethorphan; bupropion; Axsome
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label (Experimental): Experimental: AXS-05 (dextromethorphan-bupropion) up to 25 weeks
  Interventions: Drug: AXS-05 (dextromethorphan-bupropion)

INTERVENTIONS:
Drug: AXS-05 (dextromethorphan-bupropion) — AXS-05 tablets, taken twice daily

SUMMARY:
The primary objective of this open-label extension trial is to evaluate the long-term safety of AXS-05 for the treatment of Alzheimer's disease agitation in subjects that participated in ADVANCE-2 and ACCORD-2.

DETAILED DESCRIPTION:
This is a multi-center, open-label extension trial to evaluate the long-term safety of AXS-05 in subjects with Alzheimer's disease (AD) agitation that wish to continue to receive AXS-05 given completion of ADVANCE-2 (AXS-05-AD-304) and ACCORD-2 (AXS-05-AD-303).

ELIGIBILITY:
Inclusion Criteria:

* Completed the treatment period in Study AXS-05-AD-304 or exited from Study AXS-05-AD-303 due to study completion.
* Caregiver is willing to communicate with site personnel, comply with all required study procedures, and oversee administration and compliance with the subject's study treatment.

Exclusion Criteria:

* Caregiver is unwilling or unable, in the opinion of the Investigator, to comply with study instructions.
* Subject is hospitalized in a mental health facility (e.g., psychiatric hospital or ward), living in a nursing home, or living alone.
* Any concurrent medical condition that might interfere with the conduct of the study, confound the interpretation of study results, or endanger the subject's well-being.
* Initiation of a new medication since enrolling in AXS-05-AD-304 and/or AXS-05-AD-303 which may pose a safety risk when taken concurrently with AXS-05.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Long-Term Safety | Up to 25 weeks
  Incidence of treatment-emergent adverse events following dosing with AXS-05

CONTACTS AND LOCATIONS:
Locations (17):
- United States (16):
  - Clinical Research Site, Peoria, Arizona
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Bonita Springs, Florida
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Green Acres, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Gardens, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Pembroke Pines, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Braintree, Massachusetts
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, Charlotte, North Carolina
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, Arlington, Virginia
- Clinical Research Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com